CLINICAL TRIAL: NCT01883882
Title: Pilot Randomized Trial of Opioid Taper Support
Brief Title: Pilot Trial of Opioid Taper Support
Acronym: POTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Sullivan, Prinicipal Study Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 43641-B; R34DA033384 (NIH)
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Non-cancer Pain
Keywords: chronic non-cancer pain; opioid taper; chronic pain self-management; motivational interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- taper support (Experimental): Weekly visits with pharmacological and psychological support for opioid taper at 10% of original dose per week
  Interventions: Behavioral: opioid taper support
- Usual care (No Intervention): Usual care for chronic pain. All care allowed except buprenorphine.

INTERVENTIONS:
Behavioral: opioid taper support — Weekly visits with physician's assistant (supervised by pain physician/psychiatrist and pain psychologist) who provides pharmacological and psychological support for opioid taper at 10% per week
  Arms: taper support

SUMMARY:
The proposed research will develop, demonstrate the feasibility of, and pilot test in a randomized controlled trial a prescription opioid taper support intervention. This intervention aims to prevent opioid misuse and adverse events among patients receiving chronic opioid therapy for chronic non-cancer pain without evidence of current substance abuse.

The project will yield information essential to planning a future, larger-scale RCT designed to evaluate: 1) the efficacy of the intervention in preventing prescription opioid abuse, misuse, overdose and other adverse events among patients receiving chronic opioid therapy for chronic non-cancer pain, 2) the effects of the intervention on opioid use, pain, pain related activity interference, and mood. Participants in our pilot study will be limited to those without current opioid abuse or other substance abuse, but past substance abuse will be allowed. This will provide a sample of patients at risk for opioid abuse, misuse and overdose, but who may be able to taper their opioids successfully. Hypothesis: Patients receiving chronic opioid therapy for chronic non-cancer pain who are randomized to the opioid taper support intervention, as compared with patients randomized to usual opioid prescribing care, will have lower opioid average daily doses at 22 and 34 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years;
* CNCP, defined as pain on more than half the days in the past six months, where indicated diagnostic workup is complete and treatment is focused on pain;
* currently on COT, defined as self-report of prescribed oral opioid medication use on a daily or near-daily (>90% of days) basis for 90 days or more;
* mean daily opioid dose in the past 30 days of 25 mg MED or greater;
* willing to participate in the study arm to which they are randomly assigned (including opioid taper in-person sessions if randomized to that group);
* able to read, speak, and write English.

Exclusion Criteria:

* currently receiving treatment for cancer (other than non-melanoma skin cancer);
* medical comorbidity with life expectancy less than a year (based on medical record review by the PI);
* recent use (past month) of parenteral, transdermal, or transmucosal opioids,
* currently residing in nursing home;
* currently using intrathecal pump for pain control;
* any current substance abuse according to the DSM-IV checklist (nicotine and marijuana will be allowed since Washington State allows medical marijuana for pain control);
* presence of illicit drug metabolite in baseline urine drug test,
* psychotic symptoms, psychiatric hospitalization or suicide attempts in the past year;
* current suicidal ideation with specific plan or intent;
* significant cognitive impairment (on 6-item screener Scale).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-06; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
mean daily opioid dose over past week | week 22 after randomization
  mean daily opioid dose over past week as calculated in morphine equivalent dose

SECONDARY OUTCOMES:
prescription opioid difficulties | week 22 after randomization
  Prescription opioid difficulties subscale scores on: psychosocial problems and opioid control concerns

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington Center for Pain Relief, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No